CLINICAL TRIAL: NCT02191748
Title: Assessing the Efficacy of Needling With or Without Corticosteroids in the Repigmentation of Vitiligo
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Principal investigator made the decision to close study and not submit a renewal. Lack of fixed research personnel to carry out the study effectively.
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Pro2013003377
Record Dates: First submitted 2014-06-03; First posted 2014-07-16 (Estimated); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Vitiligo
MeSH Terms: conditions — Vitiligo | interventions — Triamcinolone; Triamcinolone Acetonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Needling (Active Comparator): Needling is a procedure in which a needle is inserted into normally pigmented skin on the rim of a vitiligo patch and then is pushed into the center of the patch, theoretically moving healthy, pigmented skin cells into the vitiligo patch. Saline, which doesn't affect repigmentation in vitiligo, will be injected into the patch at multiple sites spaced approximately 1 cm apart with 0.1-0.2 cc of saline injected at each site.
  Interventions: Procedure: Needling
- Needling and Triamcinolone (Experimental): During the process of needling, the needle will be attached to a syringe filled with a steroid, which is then injected into the patch, enabling delivery of the steroid directly to the affected area. Triamcinolone (concentration: 2.5 mg/cc) will be injected into the patch at multiple sites spaced approximately 1 cm apart with 0.1-0.2 cc of triamcinolone injected at each site.
  Interventions: Procedure: Needling; Drug: Triamcinolone
- No treatment (No Intervention): No treatment will be done to these vitiligo patches as a control.

INTERVENTIONS:
Procedure: Needling — Needling is a procedure in which a needle is inserted into normally pigmented skin on the rim of a vitiligo patch and then is pushed into the center of the patch, theoretically moving healthy, pigmented skin cells into the vitiligo patch.
  Arms: Needling; Needling and Triamcinolone
Drug: Triamcinolone — During the process of needling, the needle will be attached to a syringe filled with a steroid, which is then injected into the patch, enabling delivery of the steroid directly to the affected area
  Other Names: Kenalog
  Arms: Needling and Triamcinolone

SUMMARY:
Vitiligo is an autoimmune cutaneous disorder that destroys melanocytes leading to depigmented areas of skin. In the United States, vitiligo affects 1% of patients, causing not only changes in the color of skin, but also significant cosmetic concerns and quality of life issues. Current treatment modalities, which include topical corticosteroids, intralesional corticosteroids, phototherapy, and systemic immunosuppression, are variably effective in inducing repigmentation. Unfortunately, some cases of vitiligo are refractory to treatment. There is a need for new, effective modalities to treat patients with otherwise refractory vitiligo.

Needling is an office based procedure that theoretically transposes healthy, pigmented skin cells to depigmented areas using a needle in vitiligo patients. Two preliminary studies of needling as a novel treatment for vitiligo had promising results but were limited by small sample size and subjective results.

The proposed randomized control trial (RCT) will further investigate the use of needling to treat vitiligo. It differs from the previous studies in that it seeks to identify the cause of clinical benefit by comparing needling alone to needling with corticosteroid, examines a larger number of patients, and quantifies improvement using confocal microscopy. Confocal microscopy (CFM) allows non-invasive visualization of the skin on a cellular level and has been used in the past to diagnose cutaneous pigmentary conditions. This study would be the first RCT of needling in vitiligo to use an objective measure to quantify results, thus has the potential to establish needling as a novel, effective treatment for vitiligo and to evaluate the utility of CFM for monitoring response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients with 3 or more localized patches of stable vitiligo
* 2. No prior treatment or had failed previous vitiligo treatments

Exclusion Criteria:

* 1. Unstable vitiligo
* 2. Allergic to triamcinolone
* 3. Systemic treatments
* 4. Pregnancy

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2014-09; Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Repigmentation of vitiligo patch using confocal microscopy | baseline
Repigmentation of vitiligo patch using confocal microscopy | week 4 post treatment (only if repigmentation become first apparent at this time point)
Repigmentation of vitiligo patch using confocal microscopy | week 8 post treatment (only if repigmentation become first apparent at this time point
Repigmentation of vitiligo patch using confocal microscopy | week 12 post treatment (only if repigmentation become first apparent at this time point
Repigmentation of vitiligo patch using confocal microscopy | week 16 post treatment (only if repigmentation become first apparent at this time point
Repigmentation of vitiligo patch using confocal microscopy | week 20 post treatment (only if repigmentation become first apparent at this time point
Repigmentation of vitiligo patch using confocal microscopy | week 24 post treatment (only if repigmentation become first apparent at this time point
Repigmentation of vitiligo patch using confocal microscopy | week 28 post treatment

SECONDARY OUTCOMES:
Photography measure to assess repigmentation | baseline
Wood's lamp to assess repigmentation | baseline
Photography measure to assess repigmentation | week 4 post treatment
Photography measure to assess repigmentation | week 8 post treatment
Photography measure to assess repigmentation | week 12 post treatment
Photography measure to assess repigmentation | week 16 post treatment
Photography measure to assess repigmentation | week 20 post treatment
Photography measure to assess repigmentation | week 24 post treatment
Photography measure to assess repigmentation | week 28 post treatment
Wood's lamp to assess repigmentation | week 4 post treatment
Wood's lamp to assess repigmentation | week 8 post treatment
Wood's lamp to assess repigmentation | week 12 post treatment
Wood's lamp to assess repigmentation | week 16 post treatment
Wood's lamp to assess repigmentation | week 20 post treatment
Wood's lamp to assess repigmentation | week 24 post treatment
Wood's lamp to assess repigmentation | week 28 post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Babar Rao, MD, Principal Investigator — RWJUH Dermatology
Locations (1):
- RWJUH Dermatology office, Somerset, New Jersey, United States